CLINICAL TRIAL: NCT01044290
Title: Outlook: An Intervention to Improve Quality of Life in Serious Illness Study
Brief Title: Outlook Quality of Life Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIR 10-050
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Cancer; Congestive Heart Failure (CHF); Chronic Obstructive Pulmonary Disease (COPD); End Stage Renal Disease (ESRD)
Keywords: quality of life; end of life; self-disclosure; palliative care
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive; Kidney Failure, Chronic; Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Outlook Intervention (Experimental): Subjects in the first group ("Life Completion") completed a psychosocial intervention which consisted of meeting with the facilitator three times for 45-60 minutes each. In the first session, subjects were asked to discuss issues related to life review. In session two, participants spoke about issues of regret and forgiveness. In the final session, subjects focused on heritage and legacy.
  Interventions: Other: Life Completion
- Attention Control (Active Comparator): The subjects in the second group ("attention control") met with a facilitator three times for 45 minutes and listened to a non-guided relaxation CD.
  Interventions: Other: Attention Control
- Treatment as Usual (No Intervention): Subjects in the third group ("treatment as usual") were exposed to no intervention or attention control during the intervention window.

INTERVENTIONS:
Other: Life Completion — Subjects discussed life review, issues of forgiveness and heritage and legacy.
  Arms: Outlook Intervention
Other: Attention Control — Subjects listened to a non-guided relaxation CD
  Arms: Attention Control

SUMMARY:
The purpose of this study is to determine whether discussions of life story, forgiveness, and future goals improve quality of life for patients with serious illness.

DETAILED DESCRIPTION:
This is a randomized control trial to evaluate the feasibility of the Outlook intervention. 221 veterans with advanced cancer, congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD) or end stage renal disease (ESRD) were randomly assigned to one of three intervention groups and completed a brief battery of pre-test measures. Subjects in the first group ("Outlook Intervention") were randomized to meet with a facilitator three times for a period of 45 min-1 hour. Participants were asked in the first session to discuss issues related to life review. They were asked in the second session to speak in more depth about issues of regret, forgiveness and things left undone. The subject of the final session was heritage and legacy. Participants in the attention control group were randomized to meet with a facilitator three times for a period of 45 min- 1 hour and listen to a non-guided relaxation audio disc (CD). Participants in the third group ("treatment as usual") were exposed to no interventional sessions. Participants were assessed with post-test measures administered by a blinded interviewer one week and 3 weeks after the intervention window.

ELIGIBILITY:
Inclusion Criteria:

* Patients with
* Advanced cancer
* Congestive heart failure
* COPD
* End stage renal disease

Exclusion Criteria:

* Cognitive impairment
* inability to speak
* non-English speaking

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. Steinhauser, PhD, Principal Investigator — Durham VA Medical Center HSR&D COE
Locations (1):
- Durham VA Medical Center HSR&D COE, Durham, North Carolina, United States

REFERENCES:
- [Background] Steinhauser KE, Voils CI, Bosworth H, Tulsky JA. What constitutes quality of family experience at the end of life? Perspectives from family members of patients who died in the hospital. Palliat Support Care. 2015 Aug;13(4):945-52. doi: 10.1017/S1478951514000807. Epub 2014 Jul 8. PMID 25003541
- [Derived] Steinhauser KE, Alexander S, Olsen MK, Stechuchak KM, Zervakis J, Ammarell N, Byock I, Tulsky JA. Addressing Patient Emotional and Existential Needs During Serious Illness: Results of the Outlook Randomized Controlled Trial. J Pain Symptom Manage. 2017 Dec;54(6):898-908. doi: 10.1016/j.jpainsymman.2017.06.003. Epub 2017 Aug 10. PMID 28803082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 221 patients were recruited from the outpatient clinics and nursing home care unit from the Durham VA Medical Center from 1/2011 to 12/2013. Patients were eligible if they were considered to have serious life-limited disease, identified by clinical criteria, with staging/prognosis confirmed by a provider.
Pre-assignment Details: Eligible participants were consented, screened with the Mini Mental Status Exam (MMSE), given a baseline interview, then randomized to group. Reasons for not randomizing participants included death, drop-out, unable to contact, and study removal due to non-eligibility.
Groups:
- Outlook Intervention: Subjects in the first group ("Outlook Intervention") completed a psychosocial intervention which consisted of meeting with the facilitator three times for 45-60 minutes each. In the first session, subjects were asked to discuss issues related to life review. In session two, participants spoke about issues of regret and forgiveness. In the final session, subjects focused on heritage and legacy.
- Attention Control: Subjects in the second group ("attention control") met with a facilitator three times for 45 minutes and listened to a non-guided relaxation CD.
  Attention Control: Subjects will listen to a non-guided relaxation CD
- Arm 3 Treatment as Usual: Subjects in the third group ("treatment as usual") were exposed to no intervention or attention control during the intervention window.
Period: Randomization
Arm/Group | Outlook Intervention | Attention Control | Arm 3 Treatment as Usual
Started | 75 | 74 | 72
Randomized | 75 | 74 | 72
Completed | 75 | 74 | 72
Not Completed | 0 | 0 | 0
Period: Follow-up 1
Arm/Group | Outlook Intervention | Attention Control | Arm 3 Treatment as Usual
Started | 75 | 74 | 72
Completed F1 Interview | 61 | 60 | 61
Completed | 70 | 69 | 71
Not Completed | 5 | 5 | 1
Not completed — Death | 3 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 0
Period: Follow-Up 2
Arm/Group | Outlook Intervention | Attention Control | Arm 3 Treatment as Usual
Started | 70 | 69 | 71
Completed F2 Interview | 64 | 57 | 64
Completed | 70 | 67 | 69
Not Completed | 0 | 2 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: A total of 261 Durham VAMC patients with serious life-limiting disease were consented, and 221 were randomized to the study. Seventy-five were randomized to the Life completion intervention, 74 to the active control intervention, and 72 to the usual care control group.
Groups:
- Arm 1 -Outlook Intervention: Subjects in the first group ("Outlook Intervention") completed a psychosocial intervention which consists of meeting with the facilitator three times for 45-60 minutes each. In the first session, subjects were asked to discuss issues related to life review. In session two, participants spoke about issues of regret and forgiveness. In the final session, subjects focused on issues of heritage and legacy.
  Life Completion: Subjects will discuss life review, issues of forgiveness and heritage and legacy.
- Arm 2 Attention Control: The subjects in the second group ("attention control") met with a facilitator three times for 45 minutes and listen to a non-guided relaxation CD.
  Attention Control: Subjects will listen to a non-guided relaxation CD
- Total: Total of all reporting groups
Arm/Group | Arm 1 -Outlook Intervention | Arm 2 Attention Control | Arm 3 Treatment as Usual | Total
Number analyzed (Participants) | 75 | 74 | 72 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.4) | 68.2 (9.8) | 66.4 (8.3) | 67.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 68 | 70 | 212
  Male | 1 | 6 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 75 | 73 | 70 | 218
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 38 | 31 | 28 | 97
  White | 36 | 42 | 39 | 117
  More than one race | 1 | 1 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 75 | 74 | 72 | 221
Palliative Performance Scale - Stratification variable [Number; unit: participants] — The Palliative Performance Scale was used to assess functional status of participants. It was used as a stratification variable in randomization to assure that all arms of the trial had equal numbers of participants at similar levels of functional abilities, and illness severity. Scale range is 0 -100 where higher numbers indicate higher function.
  participants
    High (greater or = 70) | 55 | 55 | 54 | 164
    Low (less or = 60) | 20 | 19 | 18 | 57
Highest level of Education [Number; unit: participants]
  Less than High School (HS) degree | 6 | 7 | 8 | 21
  HS degree or GED | 25 | 29 | 25 | 79
  Some college, associate, trade school | 31 | 29 | 24 | 84
  Bachelor's degree | 8 | 4 | 9 | 21
  some graduate/professional or higher degree | 5 | 5 | 6 | 16
Religion [Number; unit: participants]
  Christian | 72 | 69 | 62 | 203
  Other | 1 | 1 | 3 | 5
  Not a member of a religion | 2 | 3 | 5 | 10
  Missing | 0 | 1 | 2 | 3
Financial Status [Number; unit: participants]
  Difficulty paying the bills | 12 | 14 | 10 | 36
  Money to pay bills but need to cut back | 20 | 19 | 19 | 58
  Pay bills but little spare money | 25 | 25 | 22 | 72
  Have enough money for special things | 18 | 16 | 21 | 55
Working Status [Number; unit: participants]
  Working for pay, part or full-time | 4 | 7 | 4 | 15
  Not working | 4 | 6 | 9 | 19
  Retired | 44 | 41 | 41 | 126
  Disability | 23 | 20 | 18 | 61

OUTCOME MEASURES:

1. Primary Outcome: QUAL-E - Preparation Sub-scale
Description: Quality Of Life At The End Of Life (the QUAL-E 2009) is a 31 item measure of quality of life at the end of life assessing five domains: life completion, relationship with health care providers, preparation for death, physical symptoms and affective social support. We include the 4-item preparation sub-scale as a primary outcomes measure. Individual items used a 5 point likert scale. The sub-scale minimum score was 5 and maximum was 20 with higher numbers indicating higher preparation.
Time Frame: Baseline (n=75, 74, 72), 5 weeks (n=61, 59, 60) and 7 weeks (n=64, 56, 64)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1 -Outlook Intervention: Participants received the Outlook Intervention
- Arm 2 Attention Control: Participants received a relaxation meditation as attention control
- Arm 3 Treatment as Usual: Participants received no intervention, but rather care as usual
Arm/Group | Arm 1 -Outlook Intervention | Arm 2 Attention Control | Arm 3 Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 72
units on a scale
  Baseline mean | 15.7 (3.3) | 14.5 (3.5) | 14.8 (3.9)
  5 week follow up | 16.0 (3.1) | 15.5 (3.3) | 14.4 (3.9)
  7 week follow up | 15.5 (3.2) | 15.2 (3.5) | 14.6 (3.5)
Statistical Analysis 1: Comparison: Arm 1 -Outlook Intervention vs Arm 2 Attention Control; Comparison at 5 weeks; Test type: Superiority or Other; p < 0.61, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = -.2, 95% CI 2-sided [-1.1 to .7]
Statistical Analysis 2: Comparison: Arm 1 -Outlook Intervention vs Arm 3 Treatment as Usual; Comparison at 5 weeks; Test type: Superiority or Other; p < .02, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = 1.1, 95% CI 2-sided [.2 to 2.0]

2. Secondary Outcome: POMS Anxiety Sub-scale
Description: The anxiety sub-scale from the modified Brief Profile of Mood States (POMS) is a 5-item measure of psychological distress.Items are on a 5-point likert scale with scoring ranging from 0-20. Higher scores indicate greater anxiety.
Time Frame: Baseline (n=75, 74, 72), 5 weeks (n=61, 60, 60), 7 weeks (n=64, 57, 64)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 2 Attention Control: Participants received a relaxation meditation as attention control condition.
- Arm 3 Treatment as Usual: Participants received no intervention but rather care as usual.
Arm/Group | Arm 1 -Outlook Intervention | Arm 2 Attention Control | Arm 3 Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 72
units on a scale
  Baseline | 5.5 (4.5) | 5.9 (4.1) | 6.5 (4.6)
  5 Weeks | 5.4 (3.8) | 5.6 (4.1) | 5.9 (4.6)
  7 Weeks | 5.9 (4.1) | 5.3 (3.8) | 6.7 (4.7)
Statistical Analysis 1: Comparison: Arm 1 -Outlook Intervention vs Arm 2 Attention Control; Comparison at 5 weeks; Test type: Superiority or Other; p = .9, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = -.1, 95% CI 2-sided [-1.2 to 1.1]
Statistical Analysis 2: Comparison: Arm 1 -Outlook Intervention vs Arm 3 Treatment as Usual; Comparison at 5 weeks; Test type: Superiority or Other; p < .97, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = -0.02, 95% CI 2-sided [-1.2 to 1.1]

3. Secondary Outcome: CES-D
Description: Center for Epidemiology Studies - Depression Scale (CES-D) is a 10-item measure of depression. Items are rated on a 4 point likert scale with total scores ranging from 0-30. Higher scores indicate greater depressive symptoms.
Time Frame: Baseline (n=75, 74, 72), 5 weeks (n=61, 60, 61) and 7 weeks (n=64, 57, 64)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 2 Attention Control: Participants received a relaxation meditation as the attention control condition.
- Arm 3 Usual Care: Participants did not receive any intervention but rather care as usual.
Arm/Group | Arm 1 -Outlook Intervention | Arm 2 Attention Control | Arm 3 Usual Care
Number analyzed (Participants) | 75 | 74 | 72
units on a scale
  Baseline | 7.9 (5.4) | 8.9 (5.8) | 9.4 (6.1)
  5 week | 8.1 (5.0) | 8.4 (5.2) | 9.2 (6.5)
  7 Week | 8.8 (5.1) | 9.2 (6.3) | 9.6 (5.5)
Statistical Analysis 1: Comparison: Arm 1 -Outlook Intervention vs Arm 2 Attention Control; Comparison at 5 weeks; Test type: Superiority or Other; p < .91, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = .1, 95% CI 2-sided [-1.4 to 1.5]
Statistical Analysis 2: Comparison: Arm 1 -Outlook Intervention vs Arm 3 Usual Care; Comparison at 5 weeks; Test type: Superiority or Other; p = .42, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.1 to 0.9]

4. Secondary Outcome: FACIT-SP
Description: The Functional Assessment of Chronic Illness Therapy- Spiritual Well-being Scale (Facit-SP) is a 12-item measure of faith, meaning and purpose, with a range of 0 to 48. Higher scores indicate greater spiritual well-being.
Time Frame: Baseline (n=75, 74, 72), 5 weeks (61, 59, 60) and 7 weeks (64, 56, 63)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 3 Treatment as Usual: Participants did not receive any intervention but rather care as usual.
Arm/Group | Arm 1 -Outlook Intervention | Arm 2 Attention Control | Arm 3 Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 72
units on a scale
  Baselin | 34.5 (8.0) | 33.6 (9.1) | 32.8 (8.8)
  5 Weeks | 34.6 (7.6) | 33.8 (8.5) | 33.9 (9.6)
  7 Weeks | 34.8 (8.0) | 34.2 (8.4) | 33.9 (9.0)
Statistical Analysis 1: Comparison: Arm 1 -Outlook Intervention vs Arm 2 Attention Control; Comparison at 5 weeks; Test type: Superiority or Other; p = .58, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = .6, 95% CI 2-sided [-1.5 to 2.8]
Statistical Analysis 2: Comparison: Arm 1 -Outlook Intervention vs Arm 3 Treatment as Usual; Comparison at 5 weeks; Test type: Superiority or Other; p < .97, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Net) = .04, 95% CI 2-sided [-2.1 to 2.2]

5. Primary Outcome: QUAL-E Life Completion Sub-scale
Description: Quality Of Life At The End Of Life (the QUAL-E 2009) is a 31 item measure of quality of life at the end of life assessing five domains: life completion, relationship with health care providers, preparation for death, physical symptoms and affective social support. We include the 7-item life completion sub-scale as a primary outcomes measure. Individual items used a 5 point likert scale. The sub-scale minimum score was 7 and maximum was 35 with higher scores indicating greater completion.
Time Frame: Baseline (n=75, 74, 72), 5 weeks (n=61, 59, 60) and 7 weeks (n=64, 55, 64)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 -Outlook Intervention | Arm 2 Attention Control | Arm 3 Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 72
units on a scale
  Baseline | 26.0 (5.3) | 26.4 (5.7) | 25.8 (5.4)
  5 weeks | 26.6 (4.6) | 26.4 (5.7) | 25.6 (6.0)
  7 weeks | 26.1 (5.1) | 27.5 (4.9) | 25.6 (4.8)
Statistical Analysis 1: Comparison: Arm 1 -Outlook Intervention vs Arm 2 Attention Control; Comparison at 5 weeks; Test type: Superiority or Other; p = .25, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Final Values) = .9, 95% CI 2-sided [-.6 to 2.4]
Statistical Analysis 2: Comparison: Arm 1 -Outlook Intervention vs Arm 3 Treatment as Usual; Comparison at 5 weeks; Test type: Superiority or Other; p < .05, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [.05 to 3.1]

6. Secondary Outcome: FACT-G - Social Sub-scale
Description: Functional assessment of Cancer Therapy-General) is a 27 item survey which assesses physical, social/family, emotional, and functional well being. This sub-scale assesses social well-being. We omitted an item assessing satisfaction with sex life, due to high missing data. Items are rated on a 5 point likert scale, with 0 indicating "not at all" and 4 indicating, "very much" in response to item questions. Total sub-scale range is 0 to 30, with higher scores indicating better well-being.
Time Frame: Baseline (n=75, 74, 72), 5 weeks (n=61, 60, 61) and 7 weeks (64, 57, 64)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 2 Attention Control: Participants received relaxation meditation as the attention control condition
Arm/Group | Arm 1 -Outlook Intervention | Arm 2 Attention Control | Arm 3 Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 72
units on a scale
  Baseline | 18.0 (4.9) | 17.4 (4.5) | 17.4 (5.1)
  5 Weeks | 18.4 (5.2) | 17.6 (4.8) | 17.1 (5.0)
  7 Weeks | 18.5 (4.6) | 18.3 (4.7) | 16.7 (5.7)
Statistical Analysis 1: Comparison: Arm 1 -Outlook Intervention vs Arm 2 Attention Control; Comparison at 5 weeks; Test type: Superiority or Other; p < .57, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable. Sex item omitted from scale; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.0 to 1.8]
Statistical Analysis 2: Comparison: Arm 1 -Outlook Intervention vs Arm 3 Treatment as Usual; Comparison at 5 weeks; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis; Adjusted for Palliative Performance Scale (low versus high) stratification variable. Sex item omitted from scale; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.03 to 2.7]

ADVERSE EVENTS:
Description: Adverse events were reported according to organ system rather than specific condition. Thus "cardiac" might include myocardial infarction as well as other cardiac events.
Groups:
- Outlook Intervention: Subjects in the first group ("Life Completion") will complete a psychosocial intervention which consists of meeting with the facilitator three times for 45-60 minutes each. In the first session, subjects will be asked to discuss issues related to life review. In session two, participants will speak about issues of regret and forgiveness. In the final session, subjects will focus on heritage and legacy.
  Life Completion: Subjects will discuss life review, issues of forgiveness and heritage and legacy.
- Attention Control: The subjects in the second group ("attention control") will meet with a facilitator three times for 45 minutes and listen to a non-guided relaxation CD.
- Treatment as Usual: Subjects in the third group ("treatment as usual") will be exposed to no intervention or attention control during the intervention window.
Arm/Group | Outlook Intervention | Attention Control | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 12/75 | 16/74 | 13/72
Other Adverse Events (participants affected / at risk) | 6/75 | 8/74 | 6/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outlook Intervention (N=75) | Attention Control (N=74) | Treatment as Usual (N=72)
cardiac (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
death (General disorders) | 3 (3) | 3 (3) | 2 (2)
general (General disorders) | 1 (1) | 3 (3) | 1 (1)
neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 1 (1)
procedural complicaton (Surgical and medical procedures) | 1 (1) | 1 (1) | 3 (3)
psychiatric (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
surgery (Surgical and medical procedures) | 2 (2) | 1 (1) | 1 (1)
respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
renal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
vascular (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outlook Intervention (N=75) | Attention Control (N=74) | Treatment as Usual (N=72)
psychiatric (Psychiatric disorders) | 3 (3) | 5 (5) | 2 (2)
infection (Infections and infestations) | 3 (3) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes